CLINICAL TRIAL: NCT00950664
Title: A Double Blind, Randomized, Multi-center, Cross-over Study to Demonstrate the Non-inferiority of Dysport® in Comparison With Botox®, Assuming a Bioequivalence Ratio of 2.5:1 Units, in the Cervical Dystonia
Brief Title: A Study to Compare Dysport® and Botox® in the Treatment of Cervical Dystonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ipsen (Industry); Medical Research Collaborating Center, Seoul, Korea (Other)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-0902-049-272
Record Dates: First submitted 2009-07-29; First posted 2009-08-03 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Cervical Dystonia
Keywords: cervical dystonia; botulinum toxin
MeSH Terms: conditions — Torticollis | interventions — abobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dysport® to Botox® (Experimental): Dysport® injection in first intervention period and Botox® in second intervention period (after washout period) cross over injection of Dysport® (abobotulinumtoxinA) and Botox® (onabotulinumtoxinA)
  Interventions: Drug: Dysport® (abobotulinumtoxinA); Drug: Botox® (onabotulinumtoxinA)
- Botox® to Dysport® (Experimental): Botox® injection in first intervention period and Dysport® in second intervention period (after washout period) cross over injection of Dysport® (abobotulinumtoxinA) and Botox® (onabotulinumtoxinA)
  Interventions: Drug: Dysport® (abobotulinumtoxinA); Drug: Botox® (onabotulinumtoxinA)

INTERVENTIONS:
Drug: Dysport® (abobotulinumtoxinA) — Cross over injection of Dysport® (<500IU), Botox® (200IU)assuming a bioequivalence ratio of 2.5:1 units
  Other Names: Dysport® (abobotulinumtoxinA)injection
Drug: Botox® (onabotulinumtoxinA) — Cross over injection of Dysport® (<500IU), Botox® (200IU)assuming a bioequivalence ratio of 2.5:1 units
  Other Names: Botox® (onabotulinumtoxinA)injection

SUMMARY:
1. to examine the non-inferiority of Dysport in the clinical efficacy and safety in comparison with Botox®, assuming a bioequivalence ratio of 2.5:1 units, in the treatment of Cervical dystonia.
2. double blind, randomised, multi center, crossover study

DETAILED DESCRIPTION:
1. Prospective, randomized, head-to-head, double-blind, cross-over study.
2. Total patients: A group 51, B group 51
3. Study duration: 16 + 4 + 16 weeks. Eligible patients will be randomised at baseline to receive either Dysport® or Botox® and monitored at weeks 2, 4, 8, 12, 16 weeks. After 4 weeks of wash out period, then the patients get the other treatment (i.e, Patients who have got Dysport will be then administered with Botox)
4. Compare the TSUI change score from baseline to 4 weeks after injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age of both genders,
* Cervical dystonia
* symptoms with a minimum duration of 18 months,
* Negative pregnancy test in sexually active women,
* Able to participate in the study (understand goals of botulinum toxin A treatment and sign Informed Consent Form).

Exclusion Criteria:

* Patient with cervical contractures
* Known significant underlying dysphasia
* Patients who have received botulinum toxin treatment within the past 4 months.
* Contraindication to botulinum toxin treatment
* Any disease that might affect neuromuscular function (Myasthenia Gravis, Eaton-Lambert syndrome, ALS …)
* Patients who have received oral anti-spasticity medication, phenol therapy, myotomy or denervation surgery, deep brain stimulation for cervical dystonia,
* Patients who required more than 500 units of Dysport or 200 units of Botox.
* Any concomitant treatment that could interfere with the action of botulinum toxin,
* Subjects having participated within the last 3 months or currently participating in an investigational drug study,
* Pregnancy,
* Lactation.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beom S Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (7):
- South Korea (7):
  - Bundang Seoul Natiuonal University Hospital, Seongnam-si, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - Hanyang University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Boramae City Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yun JY, Kim JW, Kim HT, Chung SJ, Kim JM, Cho JW, Lee JY, Lee HN, You S, Oh E, Jeong H, Kim YE, Kim HJ, Lee WY, Jeon BS. Dysport and Botox at a ratio of 2.5:1 units in cervical dystonia: a double-blind, randomized study. Mov Disord. 2015 Feb;30(2):206-13. doi: 10.1002/mds.26085. Epub 2014 Dec 5. PMID 25476727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from movement disorder clinics at 7 hospitals in Korea, between August 2009 and March 2010.
Pre-assignment Details: 103 participants recruited; 103 screened, 1 excluded (1 refused participation).
Groups:
- Dysport® First, Then Botox®: Dysport® injection in first intervention period and Botox® in second intervention period (after washout period)
- Botox® First, Then Dysport®: Botox® injection in first intervention period and Dysport® in second intervention period (after washout period)
Period: First Intervention
Arm/Group | Dysport® First, Then Botox® | Botox® First, Then Dysport®
Started | 49 | 53
Completed | 46 | 48
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 2 | 2
Period: Washout Period of 4 Weeks
Arm/Group | Dysport® First, Then Botox® | Botox® First, Then Dysport®
Started | 46 | 48
Completed | 46 | 48
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Dysport® First, Then Botox® | Botox® First, Then Dysport®
Started | 46 | 48
Completed | 0 | 0
Not Completed | 46 | 48

BASELINE CHARACTERISTICS:
Population: All analyses were performed on the modified intention-to-treat (mITT) basis, with all subjects included in the two treatment challenges.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dysport® First, Then Botox® | Botox® First, Then Dysport® | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 42 | 80
  >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.24 (11.44) | 53.35 (10.18) | 53.29 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 31 | 57
  Male | 20 | 17 | 37
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 46 | 48 | 94

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Total Tsui Score at 4 Weeks From Baseline
Description: Tsui scale is an impairment scale which evaluates the amplitude and duration of sustained posture and intermittent movements of the head, as well as the presence of shoulder elevation and tremor.
  Tsui scale (range: 0-25, higher values represent worse cervical dystonia.) Negative numbers to represent decreases of Tsui scale.
Time Frame: 4 weeks after injection from baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dysport® (abobotulinumtoxinA): Dysport® administered in either first intervention period or second intervention period
- Botox® (onabotulinumtoxinA): Botox® administered in either first intervention period or second intervention period
Arm/Group | Dysport® (abobotulinumtoxinA) | Botox® (onabotulinumtoxinA)
Number analyzed (Participants) | 94 | 94
units on a scale | -3.98 (3.89) | -4.77 (4.10)
Statistical Analysis 1: Comparison: Dysport® (abobotulinumtoxinA) vs Botox® (onabotulinumtoxinA); Test type: Non-Inferiority or Equivalence — 81 participants required to detect 5 difference in Tsui score, with 80% power. 20% drop out rate assumed, 102 participants needed. Alpha level of 0.05; p = 0.05, Paired-t test

2. Secondary Outcome: Reduction of Total TWSTRS Score at 4 Weeks From Baseline
Description: TWSTRS (Toronto western spasmodic torticollis rating scale) The TWSTRS is a composite scale which covers different features of cervical dystonia(CD).
  The first part is based on the physical findings (severity subscale), the second part rates disability, and the third part pain.
  (range: 0-80, higher values represent worse cervical dystonia.) Details of the TWSTRS are displayed on the Web site http://www.wemove.org. Negative numbers to represent decreases of TWSTRS.
Time Frame: 4 weeks after injection from baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® (abobotulinumtoxinA) | Botox® (onabotulinumtoxinA)
Number analyzed (Participants) | 94 | 94
units on a scale | -9.76 (10.25) | -8.78 (10.11)

3. Other Pre Specified Outcome: Reduction of Tsui Score at Each Visit From Baseline
Description: Tsui scale (range: 0-25, higher values represent worse cervical dystonia.) Negative numbers to represent decreases of Tsui scale.
Time Frame: 8, 12 and 16 weeks after injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® (abobotulinumtoxinA) | Botox® (onabotulinumtoxinA)
Number analyzed (Participants) | 94 | 94
units on a scale
  Reduction in Tsui Score at 8 Weeks from Baseline | -4.33 (3.69) | -4.23 (4.08)
  Reduction in Tsui Score at 12 Weeks from Baseline | -3.20 (4.48) | -3.31 (4.18)
  Reduction in Tsui Score at 16 Weeks from Baseline | -1.69 (3.99) | -1.85 (4.16)

4. Secondary Outcome: CGI-I (Clinical Global Impression of Illness)
Description: The proportion of patients with 'normal/ not at all ill' or 'borderline mildly ill' on the CGI (Clinical global impression of illness, CGI-I)
  1 = normal / not at all ill'; 2 = 'borderline mildly ill'; 3 = 'mildly ill'; 4 = 'moderlately ill'; 5 = 'markedly ill'; 6 = 'severely ill'; 7 = 'the most extremely ill'.
Time Frame: 4, 8, 12 and 16 weeks after injection
Measure: Number; unit: percentage of participants scoring 1or2
Arm/Group | Dysport® (abobotulinumtoxinA) | Botox® (onabotulinumtoxinA)
Number analyzed (Participants) | 94 | 94
percentage of participants scoring 1or2
  4 weeks after injection | 16.0 | 13.8
  8 weeks after injection | 16.0 | 14.9
  12 weeks after injection | 11.7 | 14.9
  16 weeks after injection | 8.5 | 11.7

5. Secondary Outcome: PGI-I (Patient's Global Impression of Improvement)
Description: The proportion of patients with 'very much improved' or 'much improved' on the PGI (Patient's global impression of impairment, PGI-I)
  1 = very much improved, 2= much improved, 3 = slightly improved, 4 = no change, 5 = slightly aggravated, 6 = much aggravated, and 7 = very much aggravated
Time Frame: 4, 8, 12 and 16 weeks after injection
Measure: Number; unit: percentage of patients scoring 1 or 2
Arm/Group | Dysport® (abobotulinumtoxinA) | Botox® (onabotulinumtoxinA)
Number analyzed (Participants) | 94 | 94
percentage of patients scoring 1 or 2
  4 weeks after injection | 35.1 | 36.2
  8 weeks after injection | 33.0 | 36.2
  12 weeks after injection | 20.2 | 27.7
  16 weeks after injection | 7.4 | 9.6

6. Other Pre Specified Outcome: Reduction of Total TWSTRS at Each Visit From Baseline
Description: TWSTRS scale (Toronto western spasmodic torticollis rating scale, range: 0-80, higher values represent worse cervical dystonia.) Negative numbers to represent decreases of TWSTRS scale.
Time Frame: 8, 12 and 16 weeks after injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® (abobotulinumtoxinA) | Botox® (onabotulinumtoxinA)
Number analyzed (Participants) | 94 | 94
units on a scale
  Reduction of TWSTRS from Baseline at 8 Weeks | -11.16 (10.85) | -9.98 (9.90)
  Reduction of TWSTRS from Baseline at 12 Weeks | -8.95 (11.64) | -8.66 (10.45)
  Reduction of TWSTRS from Baseline at 16 Weeks | -5.15 (8.73) | -5.34 (9.76)

7. Other Pre Specified Outcome: Reduction of Pain Associated With Cervical Dystonia at Each Visit From Baseline
Description: Pain subscale of TWSTRS scale.(Range: 0-20) Negative numbers to represent decreases of TWSTRS pain subscale.
Time Frame: 4, 8, 12 and 16 weeks after injection
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dysport® (abobotulinumtoxinA) | Botox® (onabotulinumtoxinA)
Number analyzed (Participants) | 94 | 94
units on a scale
  4 weeks after injections | -1.45 (4.05) | -1.19 (4.16)
  8 weeks after injections | -1.96 (3.97) | -2.28 (3.50)
  12 weeks after injections | -1.40 (4.08) | -2.07 (3.97)
  16 weeks after injections | -0.97 (3.85) | -1.76 (3.75)

ADVERSE EVENTS:
Time Frame: 4 Months
Arm/Group | Dysport® (abobotulinumtoxinA) | Botox® (onabotulinumtoxinA)
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/94
Other Adverse Events (participants affected / at risk) | 14/94 | 19/94
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® (abobotulinumtoxinA) (N=94) | Botox® (onabotulinumtoxinA) (N=94)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (9) | 13 (13)
Dysphagia (Musculoskeletal and connective tissue disorders) | 6 (6) | 12 (12)
Pain on neck and shoulder (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No